CLINICAL TRIAL: NCT04494152
Title: Reliability of Echocardiographic Assessment of Cardiac Dimensions and Function From Subcostal View
Brief Title: Reliability of Echocardiography From Subcostal View
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emergency Medical Service of the Central Bohemian Region, Czech Republic (Other)
Collaborators: Masaryk Hospital Usti nad Labem (Other)
Responsible Party: Principal Investigator, Roman Skulec, Principal investigator, Emergency Medical Service of the Central Bohemian Region, Czech Republic
Other Study IDs: 02/2020
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Transthoracic Echocardiography
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients: Adult critically ill patients hospitalised in the intensive care unit.
  Interventions: Diagnostic Test: Transthoracic echocardiography

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiography — Standard Point-of-Care echocardiographic examination in the intensive care unit.

SUMMARY:
The purpose of this study is to assess reliability of echocardiographic assessment of ventricular dimensions and function from subcostal view.

DETAILED DESCRIPTION:
Assessment of the function and dimensions of the right and left ventricles is a key part of Point-of-Care ultrasound in critically ill patients. According to the recent guidelines, this evaluation is performed from apical and parasternal views. However, these views may not be clearly visible in the clinical setting of critical illness and subcostal view is often preferred for its higher feasibility. Before clinical adoption, it is necessary to assess whether the isolated examination from subcostal view is reliable enough in the detection of the impairment of systolic function and the size of both ventricles and the investigators decided to evaluate this issue.

Transverse and longitudinal dimensions and function of both ventricles will be measured calculated by transthoracic echocardiography in critically ill patients in the intensive care unit from parasternal and apical views following the recent guidelines. Systolic function of the left ventricle will be expressed by the left ventricular ejection fraction (calculated by biplane method of disc summation) and by the fraction shortening. Systolic function of the right ventricle will be assessed by the tricuspid annular plane systolic excursion, fractional area change, tricuspid lateral annular systolic velocity, and right ventricular index of myocardial performance. From subcostal view, transverse dimensions of both ventricles and novel parameters of systolic function (subcostal tricuspid annular plane systolic excursion, right ventricular subcostal fraction shortening, right ventricular modified subcostal fraction shortening, left ventricular subcostal fraction shortening and left ventricular modified fraction shortening) will be measured.

Then, the reliability of parameters measured in subcostal view will be tested by comparison with conventional parameters taken from apical and parasternal view by correlation analysis and diagnostic test evaluation. The most reliable thresholds of parameters from subcostal view will be calculated by receiver operating characteristic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients
* All patients hospitalised in intensive care unit indicated for transthoracic echocardiography examination

Exclusion Criteria:

* Age <18 years
* Insufficient imaging quality of transthoracic echocardiography
* Refusal of echocardiographic examination by patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-07-28 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Reliability of left ventricular subcostal fractional shortening and left ventricular modified subcostal fractional shortening in determining the global left ventricular systolic function in critically ill patients. | During the procedure
  Left ventricular subcostal fractional shortening and left ventricular modified subcostal fractional shortening are new potential echocardiographic parameters of left ventricular systolic function measurable from subcostal view.
Reliability of right ventricular subcostal fractional shortening and right ventricular modified subcostal fractional shortening in determining the global right ventricular systolic function in critically ill patients. | During the procedure
  Right ventricular subcostal fractional shortening and right ventricular modified subcostal fractional shortening are new potential echocardiographic parameters of right ventricular systolic function measurable from subcostal view.

SECONDARY OUTCOMES:
Reliability of echocardiographic parameters evaluating the structure of the left ventricle measured in a subcostal view in critically ill patients. | During the procedure
  Quantification of the left ventricular structure (size and mass) is an important part of echocardiographic examination in critically ill patients. However, the reliability of these parameters measured in the subcostal projection has not been defined.
Reliability of echocardiographic parameters evaluating the size of the right ventricle measured in a subcostal view in critically ill patients. | During the procedure
  Quantification of the right ventricular size is an important part of echocardiographic examination in critically ill patients. However, its reliability when measured in the subcostal projection has not been defined.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Skulec, MD, PhD, Principal Investigator — Masaryk Hospital Usti nad Labem
Locations (1):
- Masaryk Hospital Usti nad Labem, Ústí nad Labem, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473